CLINICAL TRIAL: NCT03210935
Title: French National Database of Rare Dermatological Cancers: Merkel Cell Carcinoma, Inoperable or Metastatic Basal Cell Carcinoma, Cutaneous Adnexal Carcinomas
Brief Title: French National Database of Rare Dermatological Cancers
Acronym: CARADERM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: NI_2014_60
Record Dates: First submitted 2017-07-04; First posted 2017-07-07 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Adnexal Tumor of Skin; Merkel Cell Carcinoma; Advanced Basal Cell Carcinoma Requiring Systemic Treatment
Keywords: Adnexal cutaneous carcinoma; Merkel cell carcinoma; Advanced basal cell carcinoma requiring systemic treatment
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Merkel cell carcinoma
- Advanced basal cell carcinoma
- Cutaneous adnexal carcinomas

SUMMARY:
Merkel cell carcinoma, advanced basal cell carcinoma requiring systemic treatment, and cutaneous adnexal carcinomas are 3 types of rare skin cancers for which much remains unknown in terms of natural behavior, prognosis, treatment and outcomes.

CARADERM is a French prospective national cohort enrolling patients with either one of these 3 tumor types, whose objectives are :

* to provide epidemiological, clinical and socio-economic characteristics of patients
* to identify new clinical or epidemiological prognostic factors for these rare cancers
* to evaluate the impact of various treatments on outcomes

DETAILED DESCRIPTION:
CARADERM is a French national multidisciplinary project which will prospectively enroll from 37 French centers any patient presenting with Merkel cell carcinoma, advanced basal cell carcinoma requiring systemic treatment or cutaneous adnexal carcinoma.

A structured and centralized database of clinical monitoring of patients will be established. Information captured will include clinical constitutional factors, factors linked to primary carcinoma, factors linked to lymph node involvement, "American Joint Committee on Cancer" (AJCC) stage at inclusion, recurrence patterns, therapeutic interventions (medical, surgical, radiotherapy and palliative strategies) with evaluation of response, date of death, date of latest news.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed Merkel cell carcinoma, advanced basal cell carcinoma requiring systemic treatment, or cutaneous adnexal carcinoma

Exclusion Criteria:

* Subjects without Merkel cell carcinoma, advanced basal cell carcinoma requiring systemic treatment, or cutaneous adnexal carcinoma
* Patients refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed Merkel cell carcinoma, advanced basal cell carcinoma requiring systemic treatment, or cutaneous adnexal carcinoma
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2015-11-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and natural history of the 3 types of rare skin cancers | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MORTIER, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (34):
- France (34):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CH Annecy Gennevois, Annecy
  - CHU Besançon, Besançon
  - CHU Avicenne, Bobigny
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Bocage, Dijon
  - CHU de Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital La Timone, Marseille
  - Hôpital St Eloi, Montpellier
  - CHU de Nancy, Nancy
  - CHU Nantes - Place Alexis Ricordeau, Nantes
  - CHU de Nice, Nice
  - CHR d'Orleans, Orléans
  - CHU Bichat, Paris
  - CHU Cochin, Paris
  - CHU St Louis, Paris
  - CHU de Bordeaux, Pessac
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Pointe à Pitre, Pointe à Pitre
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse - Larrey, Toulouse
  - CHU de Tours, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- See also: Related Info — http://www.caraderm.org